CLINICAL TRIAL: NCT06481410
Title: Exploratory Study on the Efficacy and Safety of Methylene Blue in Treating Severe Septic Shock Patients: A Prospective, Randomized, Controlled Trial
Brief Title: Efficacy and Safety of Methylene Blue in the Treatment of Severe Septic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Yuyao People's Hospital (Other); Taizhou Enze Medical Center Group (Other); NINGBO MEDICAL CENTER LIHUIIHOSPITAI (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); The second Nanning People's Hospital (Unknown); GUI LIN PEOPLE'S HOSPITAL (Unknown); Guangxi Hospital Division of The First Affiliated Hospital, Sun Yat-sen University (Unknown); The First People's Hospital of Huzhou (Other); Hangzhou Yuhang District Second People's Hospital (Unknown); Wuming Hospital of Guangxi Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-051
Record Dates: First submitted 2024-06-21; First posted 2024-07-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock; Methylene Blue; Sepsis
Keywords: Septic Shock; Methylene blue; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, single-blind study.
Who Masked: Outcomes Assessor
Masking Description: This study implements blinding for the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene Blue Intervention Group (Experimental): Methylene blue injection, 2.5 mg/kg loading dose over 15 minutes, followed by a continuous infusion of 0.25 mg/kg/hour for 12 hours or until norepinephrine has been continuously discontinued for 4 hours, whichever comes first.
  Interventions: Drug: Methylene Blue Intervention Group
- Normal Saline Control Group (Placebo Comparator): Normal saline solution, administered in the same manner and duration as the methylene blue intervention.
  Interventions: Drug: Normal Saline Control Group

INTERVENTIONS:
Drug: Methylene Blue Intervention Group — In addition to standard treatment, patients will receive methylene blue intervention. The method is as follows: a loading dose of 2.5 mg/kg administered via micro-pump over 15 minutes, followed by a continuous infusion at a rate of 0.25 mg/kg/hour for 12 hours or until norepinephrine has been continuously discontinued for 4 hours, whichever comes first. If norepinephrine needs to be increased to 0.1 μg/kg/min before the 12-hour period ends, continue using methylene blue until the 12-hour infusion is completed.
  Arms: Methylene Blue Intervention Group
Drug: Normal Saline Control Group — In addition to standard treatment, patients will receive a placebo control with normal saline, administered for the same duration as the intervention group.
  Arms: Normal Saline Control Group

SUMMARY:
The goal of this clinical trial is to investigate whether methylene blue injection can safely and effectively improve the survival rate of patients with severe septic shock, shorten the duration of norepinephrine use, reduce the dosage of vasopressors, promptly correct hemodynamics, and improve tissue perfusion and organ function impairment.

DETAILED DESCRIPTION:
Researchers will compare methylene blue to a placebo (a look-alike substance that contains no drug) to see if methylene blue works to treat severe septic shock.

Participants will:

Administer a loading dose of 2.5 mg/kg via micro-pump over 15 minutes, followed by a maintenance infusion at a rate of 0.25 mg/kg/hour for 12 hours or until norepinephrine has been continuously discontinued for 4 hours, whichever comes first. If norepinephrine needs to be increased to 0.25 μg/kg/min before the 12-hour period ends, continue using methylene blue until the 12-hour infusion is completed.

Primary Study Endpoint

- 28-day all-cause mortality rate starting from the diagnosis of septic shock.

Secondary Study Endpoints

* Time from the start to the discontinuation of norepinephrine after the diagnosis of septic shock.
* Total dose of norepinephrine used (from enrollment to 72 hours).
* Number of days without norepinephrine within 28 days.
* Duration of mechanical ventilation.
* Rate of CRRT (Continuous Renal Replacement Therapy).
* Length of ICU stay.
* Total hospital stay.

Record the following indicators before methylene blue intervention and at 24 hours, 72 hours, and 5 days after the intervention:

* Highest serum lactate level.
* Lowest mean arterial pressure.
* Alanine aminotransferase (ALT).
* Total bilirubin.
* Creatinine.
* Oxygenation index (P/F ratio).
* Creatine kinase-MB (CK-MB).
* Troponin I (TNI).
* Systemic vascular resistance index (SVRI).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Meets the Sepsis 3.0 criteria for septic shock: patients with infection who, despite adequate fluid resuscitation, require vasopressor therapy to maintain a mean arterial pressure (MAP) of ≥ 65 mmHg and have a blood lactate concentration > 2 mmol/L.
3. Diagnosed with septic shock and started on norepinephrine within 24 hours.
4. Requires a norepinephrine dose of ≥ 0.1 μg/kg/min to maintain a MAP of ≥ 65 mmHg.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Individuals allergic to methylene blue or any components of the methylene blue injection.
3. Individuals with a personal or family history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
4. Patients with an expected survival time of less than 48 hours.
5. Patients who have been on norepinephrine for more than 24 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
28-day survival rate of enrolled patients | 28-day
  Our primary endpoint is the 28-day survival rate of enrolled patients: All enrolled patients will be followed from the time of randomization until 28 days post-enrollment, recording the survival status on the 28th day after enrollment. If a patient dies within 28 days post-enrollment, the number of survival days will be recorded.
  Note:
  1. Cases where the family requests discharge to home for end-of-life care and the patient subsequently dies will be counted as death cases.
  2. Cases where the family requests discharge for non-medical reasons such as financial constraints and no further treatment is sought will be counted as dropout cases.

SECONDARY OUTCOMES:
The duration and dosage of norepinephrine use | 28-day
  The duration of norepinephrine use：The time from the start of norepinephrine (NE) administration after sepsis diagnosis until its discontinuation. The definition of discontinuation: NE must be stopped for ≥2 hours; if NE is stopped for <2 hours, it is not considered discontinued. If NE is re-administered after being stopped for more than 2 hours, it is still considered discontinued.
  The dosage of norepinephrine use：the total dose of NE used within 72 hours after the patient is enrolled in the study.
The duration of mechanical ventilation | 28-day
  The number of days without mechanical ventilation within 28 days post-enrollment. Note: Only full days without mechanical ventilation can be counted as one day.
The duration of ICU stay | 28-day
  ICU length of stay: the number of days in the ICU starting from the time of patient enrollment in the study. Note: Some patients may have multiple ICU admissions; only the ICU stay duration after the current enrollment is recorded.
The duration of overall hospital stay | 28-day
  The duration of overall hospital stay: the total number of days hospitalized starting from the time of patient enrollment in the study. Note: Days hospitalized prior to enrollment are not included.
The safety of methylene blue injection | 28-day
  We will record the complications due to the use of methylene blue, such as hemolysis: We will determine the presence of hemolysis by daily monitoring of urine color, red blood cells, hemoglobin count in complete blood count, and bilirubin levels in liver function tests. If the patient's urine turns dark brown (similar to soy sauce), accompanied by a decrease in hemoglobin and red blood cell count and a simultaneous increase in bilirubin, hemolysis will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
You can explain the reason and contact the study initiator via email to request the data. The email address is:yuwenqiao1980@zju.edu.cn